CLINICAL TRIAL: NCT01365572
Title: Prospective, Single-blinded, Randomized Comparison of the Clinical and Angiographic Results With Intravascular Analysis of EverolimuS-Eluting Versus ZoTarolimus-Eluting steNTs for In-Stent Restenosis(ISR) Lesions: Volumetric Analysis With Intravascular Ultrasound(IVUS) : Phase IV Multicenter Trial ( RESTENT-ISR Trial )
Brief Title: New Generation Drug Eluting Stent for In-stent Restenosis of Drug Eluting Stent( RESTENT-ISR Trial )
Acronym: Restenosis
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Korea University Anam Hospital (Other)
Collaborators: Catholic Medical Center (Other); KangWon National University Hospital (Other); Kyungpook National University Hospital (Other); Kunyang University Medical center (Unknown); Kyunghee University Medical Center (Other); Kyemyeong Univerisity Medical Center (Unknown); Korea University Guro Hospital (Other); Kwandong Univerisity Medical Center (Unknown); Kwangjoo Veteran Hospital (Unknown); Eulji University (Other); Dankook University (Other); Daegoo Catholic Medical College (Unknown); Dong-A University (Other); Sejong General Hospital (Other); Busan University Medical Center (Unknown); Seoul National University Medical Center (Unknown); Sunkyungwan Univeristy Medical Center (Unknown); Suncheonyang University Medical Center (Unknown); Yonsei University (Other); Yongnam University Medical Center (Unknown); Wonkwang University Medical Center (Unknown); Inje Univerisity Medical Center (Unknown); Chonnam National University (Other); Chung-Ang University (Other); Hallym University Medical Center (Other); Chungnam National University (Other)
Responsible Party: Do-Sun Lim/ Interventional Cardiology Cardiovascular Center,, Korea University Anam Hospital
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: AN09049-004
Record Dates: First submitted 2011-05-31; First posted 2011-06-03 (Estimated); Last update posted 2011-06-03 (Estimated); Status verified 2011-03

CONDITIONS: In-stent Arterial Restenosis
Keywords: Drug-eluting stent

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Xience V, drug-eluting stent (Active Comparator): randomized implantation for DES restenotic lesion
  Interventions: Device: Xiene V stent, Endeavor Resolute stent
- Endeavor Resolute, drug-eluting stent (Active Comparator): randomized implantation for DES restenotic lesion
  Interventions: Device: Xiene V stent, Endeavor Resolute stent

INTERVENTIONS:
Device: Xiene V stent, Endeavor Resolute stent — for each lesion, randomized either Xience V stent or Endeavor Resolute stent

SUMMARY:
The purpose of this study is to evaluate the feasibility, safety, and effectiveness of EndeavorTM ResoluteTM and Xience VTM stent implantation in patients with restenosis following drug-eluting stent (DES) implantation. The investigators will evaluate clinical, angiographic and intravascular ultrasound (IVUS) assessment of 9-month efficacy of EndeavorTM ResoluteTM or Xience VTM implantation in DES restenosis and assess the vascular changes of re-treatment with DES for DES restenosis using follow-up IVUS analysis. In addition, the investigators will evaluate the effectiveness of retreatment with EndeavorTM ResoluteTM or Xience VTM stent implantation in patients with restenosis after DES

ELIGIBILITY:
Inclusion Criteria:

* In-stent restenosis (over 50% by quantitative angiographic analysis) following all types of DES; only insegment restenotic lesions without ISR are not included
* Evidence of myocardial ischemia due to restenosis (e.g., stable, unstable angina, recent infarction, silent ischemia, positive functional study or a reversible changes in the ECG with or without ischemia) or over 70% by quantitative angiographic analysis
* Repeat revascularization, needed with another stent (single stent implanted lesion, lesion length no more than 28mm )
* IVUS available lesions
* Non-emergent conditions
* Patients confirmed about study enrollment and 9 month followup angiogram and IVUS

Exclusion Criteria:

Lesion & Procedural exclusion criteria

* IVUS unavailable lesion
* Restenotic lesions following PCI of de novo lesion like as below;

  * left main lesions
  * BMS restenotic lesion
  * vein graft lesion
* Restenotic lesions following 2.25mm DES implantation
* Prior history of repeat DES implantation for DES restenosis (only conventional or cutting ballooning treatment for DES restenosis is included in this study)
* Simultaneous implantation of different types of DES on restenotic or another de novo lesions (Only same DES implantation is allowed on the restenotic or another de novo lesions)
* Patients with little possibility of performing follow-up angiogram and IVUS

General exclusion criteria

* Contraindication to anti-platelet agents & Bleeding history within prior 3 months
* Prior history or current presentation of DES thrombosis
* Age over 80 years
* Known hypersensitivity or contraindication to any of the following medications: Heparin, Aspirin, Clopidogrel, Zotarolimus, Everolimus
* Severe hepatic dysfunction (3 times normal reference values)
* Serum creatinine level over 2.0 mg/dL or end-stage renal diseases on dialysis
* LVEF less than 30%
* Pregnant women or women with potential childbearing
* An elective surgical procedure is planned that would necessitate interruption of clopidogrel during the first 9 months
* Life expectancy 1 year

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 292 (Estimated)
Dates: Start 2010-01; Primary Completion 2011-09 (Estimated); Study Completion 2012-03 (Estimated)

PRIMARY OUTCOMES:
In-stent neointimal volume index | 9 months on IVUS

SECONDARY OUTCOMES:
Major adverse cardiovascular events | 12 months
  Safety end-point; to evaluate the procedural success and the incidence of 12-month death, MI, target-vessel failure (TVF), or stent thrombosis
Efficacy end-point | 9 months
  Efficacy end-point; to evaluate the 9-month binary angiographic restenosis (≥50 percent in-stent diameter stenosis) and late loss, vascular remodeling during follow-up

CONTACTS AND LOCATIONS:
Locations (1):
- Yousei Universty Healthcare System, Seoul, South Korea